CLINICAL TRIAL: NCT06362811
Title: Assessment of Efficacy of Sacral Erector Spinae Plane Block for Postoperative Analgesia in Pediatric Rectal Biopsies: A Prospective Randomized Controlled Trial
Brief Title: Assessment of Efficacy of Sacral Erector Spinae Plane Block for Postoperative Analgesia in Pediatric Rectal Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, pinar kendigelen, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 483730
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Analgesia; Pain, Acute
Keywords: Rectal Biopsy; Sacral Erector Spinae Block
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (No Intervention): Patients will go under general anesthesia and receive only 1mcg/kg fentanyl and 10mg/kg paracetamol as analgesia intraoperatively
- General anesthesia + Sacral ESP block (Active Comparator): Patients will go under general anesthesia, receive only 1mcg/kg fentanyl and 10mg/kg paracetamol intraoperatively, and bilateral sacral ESP block
  Interventions: Procedure: Sacral Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Sacral Erector Spinae Plane Block — Ultrasound-guided bilateral injection of 1ml/kg 0.25% bupivacaine into the plane underneath the erector spinae muscles over sacral crests. The needle is inserted with in-plane technique from cranial to caudal direction over S3-4.
  Other Names: Multifidus Plane Block
  Arms: General anesthesia + Sacral ESP block

SUMMARY:
The purpose of this study is to evaluate how sacral erector spinae block changed the postoperative analgesia requirements in pediatric patients undergoing rectal biopsies under general anesthesia.

DETAILED DESCRIPTION:
Rectal biopsies in pediatric patients are performed under general anesthesia to obtain adequate tissue samples and optimize for patient comfort, well-being and safety. Post-operative pain can persist for longer than a day and requires analgesics. This study aimed to evaluate the effectiveness of sacral erector spinae block in decreasing post-operative pain scores and analgesic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing only rectal biopsy
* ASA class I-II

Exclusion Criteria:

* ASA class III or more
* Coagulation disorders
* Sacral or spinal anatomical abnormalities
* Infection around the block site
* Local anesthesia allergy

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | Postoperative 30th minute, 1st hour, 2nd hour, 4th hour, 6th hour, 12th hour and 24th hour
  Children's and Infant's Postoperative Pain Scale (CHIPPS) assessment of postoperative pain (Scores between 0 and 3 indicate no pain, and scores above 4 indicate the need for pain management.)( minimum score is 0, maximum score is 10)
Analgesia requirement | Post operative 24 hours
  If CHIPPS(Children's and Infant's Postoperative Pain Scale- minimum score is 0, maximum score is 10) score > 4, patient will receive 1mg/kg tramadol during the first post-operative hour. If CHIPPS score > 4 after 1st hour, patient will receive 10mg/kg paracetamol initially and if further assessment 30 min later is still >4 patient will receive additional 1mg/kg tramadol

SECONDARY OUTCOMES:
Complications | Post-operative 24 hours
  Presence of nausea, vomiting, apnea, hypotension, bradycardia, urinary retention and other

CONTACTS AND LOCATIONS:
Overall Officials: Ayse C Tutuncu, MD, Study Director — Istanbul University - Cerrahpasa; Pinar Kendigelen, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piraccini E, Taddei S. Sacral multifidus plane block: The correct name for sacral erector spinae plane block. J Clin Anesth. 2020 Aug;63:109754. doi: 10.1016/j.jclinane.2020.109754. Epub 2020 Feb 28. No abstract available. PMID 32120194
- [Background] Tulgar S, Senturk O, Thomas DT, Deveci U, Ozer Z. A new technique for sensory blockage of posterior branches of sacral nerves: Ultrasound guided sacral erector spinae plane block. J Clin Anesth. 2019 Nov;57:129-130. doi: 10.1016/j.jclinane.2019.04.014. Epub 2019 Apr 15. No abstract available. PMID 30999197
- [Background] Oksuz G, Arslan M, Bilal B, Gisi G, Yavuz C. Ultrasound guided sacral erector spinae block for postoperative analgesia in pediatric anoplasty surgeries. J Clin Anesth. 2020 Mar;60:88. doi: 10.1016/j.jclinane.2019.08.006. Epub 2019 Sep 3. No abstract available. PMID 31491727